CLINICAL TRIAL: NCT02066636
Title: A Phase IIIb/IV Safety Trial of Nivolumab (BMS-936558) in Subjects With Advanced or Metastatic Non-Small Cell Lung Cancer Who Have Progressed During or After Receiving At Least One Prior Systemic Regimen
Brief Title: A Safety Trial of Nivolumab in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer Who Have Progressed During or After Receiving At Least One Prior Chemotherapy Regimen
Acronym: CheckMate153
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-153
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2014-02-14; First posted 2014-02-19 (Estimated); Results first posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-09

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Nivolumab (Experimental): Nivolumab 3 mg/kg solution intravenous infusion over 30 minutes every two weeks until disease progression, unacceptable toxicity, or withdrawal of informed consent
  Interventions: Drug: Nivolumab
- Cohort B: Nivolumab (Experimental): Nivolumab 3 mg/kg solution intravenous infusion over 30 minutes every two weeks until 1 year (52 weeks).
  Discontinue treatment and at progression, retreatment allowed
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab
  Other Names: BMS-936558

SUMMARY:
The purpose of this study is to estimate the incidence and characterize the outcome of high grade, select adverse events in subjects with advanced or metastatic NSCLC treated with Nivolumab.

ELIGIBILITY:
Inclusion Criteria:

1. Target Population

* Subjects with histologically-or cytologically-documented NSCLC [squamous (SQ) or nonsquamous (NSQ)] who present with Stage IIIB/Stage IV disease (according to version 7 of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology), or with recurrent or progressive disease following multimodal therapy (radiation therapy, surgical resection or definitive chemoradiotherapy for locally advanced disease)
* Subjects must have experienced disease progression or recurrence during or after at least one systemic therapy for advanced or metastatic disease
* Each subsequent line of therapy must be preceded by disease progression. A switch of an agent within a regimen in order to manage toxicity does not define the start of a new line of therapy
* Maintenance therapy following platinum doublet-based chemotherapy is not considered as a separate regimen of therapy
* Subjects who received platinum-containing adjuvant, neoadjuvant or definitive chemoradiation therapy given for locally advanced disease, and developed recurrent (local or metastatic) disease within 6 months of completing therapy are eligible
* Subjects with recurrent disease >6 months after platinum-containing adjuvant, neoadjuvant or definitive chemoradiation therapy given for locally advanced disease, who also subsequently progressed during or after a platinum doublet-based regimen given to treat the recurrence are eligible
* Subjects with non-squamous histology must be tested for Epithelial Growth Factor Receptor (EGFR) mutations (including, but not limited to, deletions in exon 19 and exon 21 [L858R] substitution) and Anaplastic Lymphoma Kinase (ALK) rearrangement if tests have not been previously performed. Subjects with progressive disease during or after EGFR or ALK tyrosine kinase inhibitor (TKI) regimens are eligible. Subjects are eligible if genetic test results are indeterminate or if no tumor tissue is available or accessible for testing as long as they have received one prior systemic therapy
* Experimental therapies when given as separate regimen are considered as separate line of therapy
* Subjects must have measurable disease by CT or MRI per RECIST 1.1 criteria (radiographic tumor assessment performed within 28 days of first dose of study drug) or clinically apparent disease that the investigator can follow for response per RECIST 1.1
* Eastern Cooperative Oncology Arm (ECOG) performance status (PS)
* PS 0 to 1
* PS 2

Exclusion Criteria:

1. Target Disease Exceptions

   * Subjects with active central nervous system (CNS) metastases are excluded
   * Subjects with carcinomatous meningitis
2. Medical History and Concurrent Diseases

   * Subjects with a history of interstitial lung disease
   * Subjects with active, known or suspected autoimmune disease
   * Subject whom participated in either arm of the following clinical trials CA209-017, CA209-057, CA209-026, and CA184-104 or received prior treatment with anti-programmed death 1 (PD-1) or anti-programmed death-ligand 1 (PDL1) experimental agents
3. Prohibited Treatments and/or Restricted Therapies

   * Ongoing or planned administration of anti-cancer therapies other than those specified in this study
   * Use of corticosteroids or other immunosuppressive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1428 (Actual)
Dates: Start 2014-04-09 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (133):
- United States (126):
  - Southern Cancer Center Pc, Mobile, Alabama
  - Cancer Center Treatment Center of America, Goodyear, Arizona
  - Arizona Oncology Associates, Phoenix, Arizona
  - Arizona Oncology Associates, Sedona, Arizona
  - Arizona Oncol Assoc Dba (Hem Onc Physicians&Extenders) Hope, Tucson, Arizona
  - Comprehensive Blood And Cancer Center, Bakersfield, California
  - Diablo Valley Oncology, Concord, California
  - Saint Jude Heritage Medical Group Virginia K Crosson Cancer Center, Fullerton, California
  - Ucla Hema/Onc-Santa Monica, Los Angeles, California
  - Pacific Cancer Care, Monterey, California
  - Sutter Cancer Center, Sacramento, California
  - Local Institution, San Francisco, California
  - Central Coast Med Oncology, San Luis Obispo, California
  - Sansum Santa Barbara Medical Foundation Clinic, Santa Barbara, California
  - Central Coast Med Oncology, Santa Maria, California
  - Torrance Memorial Medical Center, Torrance, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - St. Mary's Hospital Regional Cancer Center, Grand Junction, Colorado
  - Eastern Ct Hem Onc Assoc, Norwich, Connecticut
  - Holy Cross Hospital Inc., Fort Lauderdale, Florida
  - Florida Cancer Specialists S., Fort Myers, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Local Institution - 0031, Lakeland, Florida
  - Local Institution - 0038, Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Cancer Institute Of Florida, Orlando, Florida
  - Memorial Cancer Institute, Pemroke Pines, Florida
  - Local Institution - 0071, Pensacola, Florida
  - Hematology/Oncology Associates Of The Treasure Coast, Port Saint Lucie, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Local Institution - 0108, Tampa, Florida
  - Space Coast Cancer Center, Titusville, Florida
  - University Cancer Blood Ctr, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Central Georgia Cancer Care, Pc, Macon, Georgia
  - Cancer Treatment Centers Of America, Newnan, Georgia
  - Summit Cancer Care, Savannah, Georgia
  - Lewis Hall Singletary Oncology Center, Thomasville, Georgia
  - Pearlman Cancer Center, Valdosta, Georgia
  - University Of Illinois Cancer Center, Chicago, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Oncology Specialists, Park Ridge, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Local Institution - 0015, Skokie, Illinois
  - Southern Illinois University School Of Medicine, Springfield, Illinois
  - Local Institution - 0081, Fort Wayne, Indiana
  - Indiana University Health Melvin And Bren Simon Cancer Center, Indianapolis, Indiana
  - Cancer Center Of Kansas, Wichita, Kansas
  - Norton Cancer Center, Louisville, Kentucky
  - University Medical Center, Inc, Louisville, Kentucky
  - West KY Hematology Oncology Group PSC, Paducah, Kentucky
  - Christus Schumpert Health, Shreveport, Louisiana
  - Local Institution, Brewer, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Walter Reed National Mltry Medical Center, Bethesda, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Bay Hematology Oncology, Easton, Maryland
  - Michigan Cancer Research Consortinum, Ann Arbor, Michigan
  - Cancer & Hematology Centers Of Western Michigan, Grand Rapids, Michigan
  - Providence Cancer Center, Southfield, Michigan
  - Forrest General Cancer Center, Hattiesburg, Mississippi
  - Jackson Oncology Associates, Pllc, Jackson, Mississippi
  - North Mississippi Hematology And Oncology Associates, Ltd, Tupelo, Mississippi
  - University Of Kansas Cancer Center, North Kansas City, Missouri
  - Mercy Medical Research Institute, Springfield, Missouri
  - Southeast Nebraska Hematology & Oncology Consultants, P.C., Lincoln, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Center Of Nevada, Las Vegas, Nevada
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - Hunterdon Medical Center, Flemington, New Jersey
  - Atlantic Health System, Summit, New Jersey
  - Presbyterian Medical Group, Albuquerque, New Mexico
  - St. Peters Hospital, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Queens Medical Associates, Fresh Meadows, New York
  - Broome Oncology, Johnson City, New York
  - Winthrop University Hospital, Mineola, New York
  - Mount Kisco Medical Group, Mount Kisco, New York
  - Columbia University Medical Center (Cumc), New York, New York
  - Hematology-Oncology Associates Of Rockland, Nyack, New York
  - Randolph Cancer Center, Asheboro, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center, Greensboro, North Carolina
  - East Carolina University Leo W. Jenkins Cancer Center, Greeville, North Carolina
  - W.G. Bill Hefner VA Medical Center, Salisbury, North Carolina
  - Mid Dakota Clinic, Pc, Bismarck, North Dakota
  - Oncology Hematology Care, Incorporated, Cincinnati, Ohio
  - Local Institution, Cleveland, Ohio
  - Zangmeister Cancer Center, Columbus, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's University Hospital Bethlehem, Bethlehem, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology Associates, Pa, Charleston, South Carolina
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Tennessee Oncology, PLLC - SCRI - PPDS, Chattanooga, Tennessee
  - Cancer Care Of Wnc, Germantown, Tennessee
  - The Jones Clinic, PC, Germantown, Tennessee
  - The West Clinic, P.C., Germantown, Tennessee
  - Tennessee Oncology, Pllc, Nashville, Tennessee
  - Henry-Joyce Cancer Center, Nashville, Tennessee
  - Texas Oncology-Abilene, Abilene, Texas
  - Texas Oncology - Amarillo, Amarillo, Texas
  - Texas Oncology, Arlington, Texas
  - Texas Oncology-Beaumont, Beaumont, Texas
  - Texas Oncology, Bedford, Texas
  - Texas Oncology, Dallas, Texas
  - Local Institution - 0067, Dallas, Texas
  - Texas Oncology, Denton, Texas
  - The Center For Cancer And Blood Disorders, Fort Worth, Texas
  - Northwest Cancer Center, Houston, Texas
  - Texas Oncology, McAllen, Texas
  - Texas Oncology, Mesquite, Texas
  - Texas Oncology - Odessa, Midland, Texas
  - Texas Oncology-Plano East, Plano, Texas
  - Cancer Care Centers Of South Texas, San Antonio, Texas
  - Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology Cancer Care And Research Center, Waco, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University Of Virginia Health System., Charlottesville, Virginia
  - Shenandoah Oncology, Winchester, Virginia
- Canada (7):
  - Local Institution, Calgary, Alberta
  - Local Institution, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Lévis, Quebec
  - Local Institution, Montreal, Quebec

REFERENCES:
- [Derived] Spigel DR, McCleod M, Jotte RM, Einhorn L, Horn L, Waterhouse DM, Creelan B, Babu S, Leighl NB, Chandler JC, Couture F, Keogh G, Goss G, Daniel DB, Garon EB, Schwartzberg LS, Sen R, Korytowsky B, Li A, Aanur N, Hussein MA. Safety, Efficacy, and Patient-Reported Health-Related Quality of Life and Symptom Burden with Nivolumab in Patients with Advanced Non-Small Cell Lung Cancer, Including Patients Aged 70 Years or Older or with Poor Performance Status (CheckMate 153). J Thorac Oncol. 2019 Sep;14(9):1628-1639. doi: 10.1016/j.jtho.2019.05.010. Epub 2019 May 20. PMID 31121324
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After 1 year of treatment, participants who are still on treatment are randomized to Cohort A or Cohort B.
Groups:
- Cohort A: Nivolumab Monotherapy: Participants receive nivolumab administered intravenously at 3 mg/kg every two weeks. Each 14 day dosing period will constitute a cycle. After 1 year (52 weeks) of treatment all participants will continue to receive treatment until disease progression, unacceptable toxicity, or withdrawal of informed consent.
- Cohort B: Nivolumab Monotherapy: Participants receive nivolumab administered intravenously at 3 mg/kg every two weeks. Each 14 day dosing period will constitute a cycle. After 1 year (52 weeks) of treatment all participants will discontinue treatment. Upon progression, participants can receive retreatment.
- Nivolumab Monotherapy (Not Randomized): Participants receive nivolumab administered intravenously at 3 mg/kg every two weeks. Non-randomized participants were those participants who were enrolled but (after 1 year) were not randomized to either of the study cohorts (Cohort A or B).
Period: Overall Study
Arm/Group | Cohort A: Nivolumab Monotherapy | Cohort B: Nivolumab Monotherapy | Nivolumab Monotherapy (Not Randomized)
Started | 127 | 125 | 1176
Completed | 0 | 0 | 0
Not Completed | 127 | 125 | 1176
Not completed — Disease progression | 51 | 60 | 700
Not completed — Study drug toxicity | 13 | 2 | 58
Not completed — Death | 4 | 2 | 158
Not completed — Adverse event unrelated to study drug | 6 | 4 | 45
Not completed — Participant request to discontinue treatment | 12 | 12 | 70
Not completed — Participant withdrew consent | 10 | 18 | 61
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Maximum clinical benefit | 2 | 2 | 3
Not completed — Poor/non-compliance | 2 | 1 | 1
Not completed — Participant no loner meets study criteria | 3 | 2 | 28
Not completed — Administrative reasons by sponsor | 8 | 5 | 0
Not completed — Other reasons | 16 | 15 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Nivolumab Monotherapy | Cohort B: Nivolumab Monotherapy | Nivolumab Monotherapy (Not Randomized) | Total
Number analyzed (Participants) | 127 | 125 | 1176 | 1428
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (10.27) | 66.6 (7.97) | 66.1 (9.82) | 66.1 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 62 | 528 | 657
  Male | 60 | 63 | 648 | 771
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 31 | 41
  Not Hispanic or Latino | 124 | 118 | 1139 | 1381
  Unknown or Not Reported | 0 | 0 | 6 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 4 | 5
  Asian | 3 | 1 | 38 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
  Black or African American | 13 | 8 | 84 | 105
  White | 111 | 114 | 1041 | 1266
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 7 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Treatment Related Select Adverse Events (Grade 3-4 and Grade 5)
Description: A treatment related adverse event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered an investigational (medicinal) product and that has a causal relationship with this treatment. The select AEs categories are those that are expected to be most commonly used to describe pneumonitis, interstitial nephritis, diarrhea/colitis, hepatitis, rash, and endocrinopathies and hypersensitivity/infusion reactions. AEs are graded according to NCI CTCAE (Version 4.0) guidelines where Grade 3= Severe, Grade 4 = Life-threatening, Grade 5 = Death.
Time Frame: From first dose and 100 days after last dose (last dose up to randomization for cohort B) (up to approximately 88 months)
Population: All treated participants prior to randomization and treated participants randomized to Cohort A and B
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Nivolumab Monotherapy (Post-Randomization): All participants that continued to receive treatment after completing 1 year (52 weeks) of nivolumab administered intravenously at 3 mg/kg every two weeks until disease progression, unacceptable toxicity, or withdrawal of informed consent.
- Cohort B: Nivolumab Monotherapy (Post-Randomization): All participants that discontinued treatment after 1 year (52 weeks) of receiving nivolumab administered intravenously at 3 mg/kg every two weeks. Upon progression, participants can receive retreatment.
- Nivolumab Monotherapy (Pre-Randomized): All Participants that received nivolumab administered intravenously at 3 mg/kg every two weeks for up to 1 year.
Arm/Group | Cohort A: Nivolumab Monotherapy (Post-Randomization) | Cohort B: Nivolumab Monotherapy (Post-Randomization) | Nivolumab Monotherapy (Pre-Randomized)
Number analyzed (Participants) | 127 | 125 | 1428
Participants
  Gastrointestinal Adverse Event (Grade3-4) | 3 | 0 | 20
  Gastrointestinal Adverse Event (Grade 5) | 0 | 0 | 1
  Hepatic Adverse Event (Grade3-4) | 1 | 0 | 19
  Hepatic Adverse Event (Grade 5) | 0 | 0 | 0
  Pulmonary Adverse Event (Grade3-4) | 1 | 1 | 18
  Pulmonary Adverse Event (Grade 5) | 0 | 0 | 0
  Renal Adverse Event (Grade3-4) | 0 | 0 | 4
  Renal Adverse Event (Grade 5) | 0 | 0 | 0
  Skin Adverse Event (Grade3-4) | 1 | 1 | 15
  Skin Adverse Event (Grade 5) | 0 | 0 | 0
  Hypersensitivity/Infusion Reaction Events (Grade3-4) | 0 | 0 | 4
  Hypersensitivity/Infusion Reaction Events (Grade 5) | 0 | 0 | 0
  Endocrinopathies (Grade3-4) | 0 | 0 | 6
  Endocrinopathies (Grade 5) | 0 | 0 | 0

2. Secondary Outcome: Median Time to Onset of Select Adverse Events (Grade 3-5)
Description: The time from first dose to the first occurrence of any select adverse event of interest. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. The select AEs categories are those that are expected to be most commonly used to describe pneumonitis, interstitial nephritis, diarrhea/colitis, hepatitis, rash, and endocrinopathies and hypersensitivity/infusion reactions. AEs are graded according to NCI CTCAE (Version 4.0) guidelines where Grade 3= Severe, Grade 4 = Life-threatening, Grade 5 = Death.
Time Frame: as for outcome 1
Population: All treated participants (both included and excluded from Cohort randomization) with at least one select adverse event from the category
Measure: Median (Full Range); unit: Weeks
Arm/Group | Cohort A: Nivolumab Monotherapy (Post-Randomization) | Cohort B: Nivolumab Monotherapy (Post-Randomization) | Nivolumab Monotherapy (Not Randomized)
Number analyzed (Participants) | 10 | 4 | 38
Weeks
  Endocrine Adverse Event: number analyzed (Participants) | 3 | 1 | 3
  Endocrine Adverse Event | 12.14 [11.0 to 45.4] | 25.3 [25.3 to 25.3] | 11.14 [5.6 to 42.7]
  Gastrointestinal Adverse Event: number analyzed (Participants) | 10 | 4 | 29
  Gastrointestinal Adverse Event | 82.71 [22.7 to 272.3] | 49.21 [33.9 to 59.4] | 17.86 [0.7 to 46.1]
  Hepatic Adverse Event: number analyzed (Participants) | 2 | 0 | 33
  Hepatic Adverse Event | 84.50 [16.4 to 152.6] |  | 4.14 [1.3 to 42.1]
  Pulmonary Adverse Event: number analyzed (Participants) | 2 | 0 | 38
  Pulmonary Adverse Event | 156.21 [97.9 to 214.6] |  | 7.79 [0.6 to 35.9]
  Renal Adverse Event: number analyzed (Participants) | 2 | 1 | 13
  Renal Adverse Event | 108.00 [35.9 to 180.1] | 15.1 [15.1 to 15.1] | 6.71 [3.0 to 49.6]
  Skin Adverse Event: number analyzed (Participants) | 5 | 2 | 11
  Skin Adverse Event | 26.14 [0.1 to 48.1] | 18.14 [16.1 to 20.1] | 10.57 [2.1 to 51.6]
  Hypersensitivity/Infusion Reaction: number analyzed (Participants) | 0 | 1 | 4
  Hypersensitivity/Infusion Reaction |  | 42.00 [42.0 to 42.0] | 2.36 [2.0 to 8.1]

3. Secondary Outcome: Median Time to Resolution of Select Adverse Events (Grade 3-5)
Description: The time from the onset of any select adverse event of interest to its resolution or stabilization. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. The select AEs categories are those that are expected to be most commonly used to describe pneumonitis, interstitial nephritis, diarrhea/colitis, hepatitis, rash, and endocrinopathies and hypersensitivity/infusion reactions. AEs are graded according to NCI CTCAE (Version 4.0) guidelines where Grade 3= Severe, Grade 4 = Life-threatening, Grade 5 = Death.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Weeks
Arm/Group | Cohort A: Nivolumab Monotherapy (Post-Randomization) | Cohort B: Nivolumab Monotherapy (Post-Randomization) | Nivolumab Monotherapy (Not Randomized)
Number analyzed (Participants) | 10 | 4 | 38
Weeks
  Endocrine Adverse Event: number analyzed (Participants) | 3 | 1 | 3
  Endocrine Adverse Event | 3.43 [0.4 to 36.1] | 1.00 [1.0 to 1.0] | 3.57 [0.9 to 4.4]
  Gastrointestinal Adverse Event: number analyzed (Participants) | 10 | 4 | 29
  Gastrointestinal Adverse Event | 4.79 [0.4 to 29.4] | 1.50 [0.3 to 3.0] | 1.86 [0.6 to 27.1]
  Hepatic Adverse Event: number analyzed (Participants) | 2 | 0 | 33
  Hepatic Adverse Event | 1.36 [0.4 to 2.3] |  | 12.57 [0.1 to 36.9]
  Pulmonary Adverse Event: number analyzed (Participants) | 2 | 0 | 38
  Pulmonary Adverse Event | 1.14 [0.7 to 1.6] |  | 2.57 [0.1 to 30.3]
  Renal Adverse Event: number analyzed (Participants) | 2 | 1 | 13
  Renal Adverse Event | 0.64 [0.4 to 0.9] | 1.9 [1.9 to 1.9] | 1.29 [0.3 to 5.1]
  Skin Adverse Event: number analyzed (Participants) | 5 | 2 | 11
  Skin Adverse Event | 2.57 [2.1 to 32.9] | 2.43 [2.1 to 2.7] | 9.14 [1.0 to 234]
  Hypersensitivity/Infusion Reaction: number analyzed (Participants) | 0 | 1 | 4
  Hypersensitivity/Infusion Reaction |  | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1]

4. Secondary Outcome: The Number of Participants Who Received Immune Modulating Medication (or Hormonal Replacement Therapy) for Any Grade Select Adverse Events
Description: The number of participants receiving medication meant to trigger an immune response for any select Adverse events of interest. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. The select AEs categories are those that are expected to be most commonly used to describe pneumonitis, interstitial nephritis, diarrhea/colitis, hepatitis, rash, and endocrinopathies and hypersensitivity/infusion reactions. AEs are graded according to NCI CTCAE (Version 4.0) guidelines where Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4 = Life-threatening, Grade 5 = Death.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab Monotherapy (Post-Randomization) | Cohort B: Nivolumab Monotherapy (Post-Randomization) | Nivolumab Monotherapy (Not Randomized)
Number analyzed (Participants) | 40 | 17 | 314
Participants
  Endocrine Adverse Event: number analyzed (Participants) | 12 | 9 | 209
  Endocrine Adverse Event | 1 | 2 | 15
  Gastrointestinal Adverse Event: number analyzed (Participants) | 40 | 17 | 288
  Gastrointestinal Adverse Event | 5 | 2 | 35
  Hepatic Adverse Event: number analyzed (Participants) | 7 | 6 | 122
  Hepatic Adverse Event | 0 | 0 | 13
  Pulmonary Adverse Event: number analyzed (Participants) | 12 | 6 | 73
  Pulmonary Adverse Event | 11 | 4 | 42
  Renal Adverse Event: number analyzed (Participants) | 21 | 5 | 96
  Renal Adverse Event | 1 | 0 | 12
  Skin Adverse Event: number analyzed (Participants) | 33 | 16 | 314
  Skin Adverse Event | 17 | 8 | 113
  Hypersensitivity/Infusion Reaction: number analyzed (Participants) | 2 | 2 | 33
  Hypersensitivity/Infusion Reaction | 2 | 1 | 14

5. Secondary Outcome: The Number of Participants Who Received ≥ 40 mg Prednisone Equivalents for Any Grade Select Adverse Events
Description: The number of participants receiving > 40mg prednisone equivalents for any select adverse event of interest. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. The select AEs categories are those that are expected to be most commonly used to describe pneumonitis, interstitial nephritis, diarrhea/colitis, hepatitis, rash, and endocrinopathies and hypersensitivity/infusion reactions. AEs are graded according to NCI CTCAE (Version 4.0) guidelines where Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4 = Life-threatening, Grade 5 = Death.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab Monotherapy (Post-Randomization) | Cohort B: Nivolumab Monotherapy (Post-Randomization) | Nivolumab Monotherapy (Not Randomized)
Number analyzed (Participants) | 40 | 17 | 314
Participants
  Endocrine Adverse Event: number analyzed (Participants) | 12 | 9 | 209
  Endocrine Adverse Event | 0 | 0 | 5
  Gastrointestinal Adverse Event: number analyzed (Participants) | 40 | 17 | 288
  Gastrointestinal Adverse Event | 3 | 2 | 21
  Hepatic Adverse Event: number analyzed (Participants) | 7 | 6 | 122
  Hepatic Adverse Event | 0 | 0 | 8
  Pulmonary Adverse Event: number analyzed (Participants) | 12 | 6 | 73
  Pulmonary Adverse Event | 7 | 4 | 31
  Renal Adverse Event: number analyzed (Participants) | 21 | 5 | 96
  Renal Adverse Event | 1 | 0 | 10
  Skin Adverse Event: number analyzed (Participants) | 33 | 16 | 314
  Skin Adverse Event | 2 | 2 | 14
  Hypersensitivity/Infusion Reaction: number analyzed (Participants) | 2 | 2 | 33
  Hypersensitivity/Infusion Reaction | 2 | 1 | 3

6. Secondary Outcome: The Total Duration of All Immune Modulating Medications for Any Grade Select Adverse Events
Description: The duration of time participants received medication meant to trigger an immune response for any select Adverse events of interest. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. The select AEs categories are those that are expected to be most commonly used to describe pneumonitis, interstitial nephritis, diarrhea/colitis, hepatitis, rash, and endocrinopathies and hypersensitivity/infusion reactions. AEs are graded according to NCI CTCAE (Version 4.0) guidelines where Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4 = Life-threatening, Grade 5 = Death.
Time Frame: From first dose first dose and 100 days after last dose (last dose up to randomization for cohort B) (up to approximately 88 months)
Population: as for outcome 2
Measure: Median (Full Range); unit: Weeks
Arm/Group | Cohort A: Nivolumab Monotherapy (Post-Randomization) | Cohort B: Nivolumab Monotherapy (Post-Randomization) | Nivolumab Monotherapy (Not Randomized)
Number analyzed (Participants) | 40 | 17 | 314
Weeks
  Endocrine Adverse Event: number analyzed (Participants) | 12 | 9 | 209
  Endocrine Adverse Event | NA [NA to NA] — Insufficient number of participants with events | 82.57 [2.0 to 163.1] | 2.57 [0.1 to 76.0]
  Gastrointestinal Adverse Event: number analyzed (Participants) | 40 | 17 | 288
  Gastrointestinal Adverse Event | 5.43 [2.4 to 8.1] | 2.50 [1.6 to 3.4] | 3.79 [0.4 to 32.6]
  Hepatic Adverse Event: number analyzed (Participants) | 7 | 6 | 122
  Hepatic Adverse Event | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | 5.0 [0.4 to 14.0]
  Pulmonary Adverse Event: number analyzed (Participants) | 12 | 6 | 73
  Pulmonary Adverse Event | 6.57 [0.3 to 27.1] | 2.86 [1.1 to 5.9] | 3.57 [0.1 to 26.1]
  Renal Adverse Event: number analyzed (Participants) | 21 | 5 | 96
  Renal Adverse Event | 0.7 [0.7 to 0.7] | NA [NA to NA] — Insufficient number of participants with events | 2.57 [0.3 to 16.9]
  Skin Adverse Event: number analyzed (Participants) | 33 | 16 | 314
  Skin Adverse Event | 18.14 [0.9 to 151.0] | 6.71 [1.0 to 16.4] | 4.07 [0.1 to 80.1]
  Hypersensitivity/Infusion Reaction: number analyzed (Participants) | 2 | 2 | 33
  Hypersensitivity/Infusion Reaction | 2.71 [1.0 to 4.4] | 2.0 [2.0 to 2.0] | 0.14 [0.1 to 2.1]

7. Secondary Outcome: The Number of Participants With High Grade (Grade 3-4 and Grade 5) Select Adverse Events
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. The select AEs categories are those that are expected to be most commonly used to describe pneumonitis, interstitial nephritis, diarrhea/colitis, hepatitis, rash, and endocrinopathies and hypersensitivity/infusion reactions. AEs are graded according to NCI CTCAE (Version 4.0) guidelines where Grade 3= Severe, Grade 4 = Life-threatening, Grade 5 = Death.
Time Frame: as for outcome 1
Population: All treated participants prior to randomization and treated participants randomized to Cohort A and B
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Nivolumab Monotherapy (Post-Randomization) | Cohort B: Nivolumab Monotherapy (Post-Randomization) | Nivolumab Monotherapy (Pre-Randomized)
Number analyzed (Participants) | 127 | 125 | 1428
Participants
  Gastrointestinal Adverse Event (Grade3-4) | 7 | 2 | 35
  Gastrointestinal Adverse Event (Grade 5) | 0 | 0 | 1
  Hepatic Adverse Event (Grade3-4) | 1 | 0 | 34
  Hepatic Adverse Event (Grade 5) | 0 | 0 | 0
  Pulmonary Adverse Event (Grade3-4) | 2 | 3 | 31
  Pulmonary Adverse Event (Grade 5) | 0 | 0 | 7
  Renal Adverse Event (Grade3-4) | 1 | 1 | 14
  Renal Adverse Event (Grade 5) | 0 | 0 | 1
  Skin Adverse Event (Grade3-4) | 1 | 2 | 18
  Skin Adverse Event (Grade 5) | 0 | 0 | 0
  Hypersensitivity/Infusion Reaction Events (Grade3-4) | 0 | 0 | 5
  Hypersensitivity/Infusion Reaction Events (Grade 5) | 0 | 0 | 0
  Endocrinopathies (Grade3-4) | 0 | 0 | 8
  Endocrinopathies (Grade 5) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to study completion (up to approximately 90 months) . SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 88 months).
Description: Post-Randomization indicates only data after randomization is summarized (applies to Cohort A and B). Pre-Randomized indicates only data before randomization is summarized (applies to all treated participants). Total indicates data is summarized throughout the full duration of the study (applies to all treated participants).
Groups:
- Nivolumab Monotherapy (Total): All Participants that received nivolumab administered intravenously at 3 mg/kg every two weeks regardless of continuation or discontinuation of treatment.
Arm/Group | Cohort A: Nivolumab Monotherapy (Post-Randomization) | Cohort B: Nivolumab Monotherapy (Post-Randomization) | Nivolumab Monotherapy (Pre-Randomized) | Nivolumab Monotherapy (Total)
All-Cause Mortality (participants affected / at risk) | 63/127 | 77/125 | 1040/1428 | 1180/1428
Serious Adverse Events (participants affected / at risk) | 57/127 | 52/125 | 870/1428 | 918/1428
Other Adverse Events (participants affected / at risk) | 101/127 | 82/125 | 1287/1428 | 1306/1428
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Nivolumab Monotherapy (Post-Randomization) (N=127) | Cohort B: Nivolumab Monotherapy (Post-Randomization) (N=125) | Nivolumab Monotherapy (Pre-Randomized) (N=1428) | Nivolumab Monotherapy (Total) (N=1428)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 12 | 13
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 7 | 7
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 5
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 5 | 5
Angina pectoris (Cardiac disorders) | 0 | 1 | 2 | 2
Angina unstable (Cardiac disorders) | 1 | 0 | 1 | 2
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 12 | 14
Atrial flutter (Cardiac disorders) | 1 | 0 | 2 | 3
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 1 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 4 | 5
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 3 | 4
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 9 | 10
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 6 | 7
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 7 | 8
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 2
Pericardial effusion (Cardiac disorders) | 1 | 0 | 11 | 12
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 2 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 5 | 5
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 2
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 2 | 2
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 0 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 1
Ocular myasthenia (Eye disorders) | 0 | 0 | 1 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 17 | 18
Colitis (Gastrointestinal disorders) | 4 | 0 | 7 | 10
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 8 | 8
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 13 | 14
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 8 | 8
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Enterocolonic fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 3 | 5
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 6 | 6
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 3 | 3
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 4 | 4
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 12 | 13
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Oesophageal fistula (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 4 | 5
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 9 | 10
Asthenia (General disorders) | 0 | 0 | 8 | 8
Catheter site injury (General disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 4 | 4
Death (General disorders) | 0 | 0 | 14 | 14
Fatigue (General disorders) | 0 | 0 | 9 | 9
General physical health deterioration (General disorders) | 0 | 0 | 2 | 2
Generalised oedema (General disorders) | 0 | 0 | 1 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 1 | 1
Localised oedema (General disorders) | 0 | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 15 | 15
Oedema peripheral (General disorders) | 0 | 0 | 2 | 2
Pain (General disorders) | 0 | 0 | 3 | 3
Physical deconditioning (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 2 | 8 | 8
Sudden death (General disorders) | 1 | 0 | 2 | 3
Autoimmune cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 3 | 3
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 3 | 3
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 3 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 1
Abscess intestinal (Infections and infestations) | 0 | 0 | 2 | 2
Abscess oral (Infections and infestations) | 0 | 0 | 1 | 1
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 3 | 3
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 2 | 1 | 4 | 6
Catheter site cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 3 | 4
Clostridium difficile colitis (Infections and infestations) | 2 | 0 | 0 | 2
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 1 | 1
Cryptococcosis (Infections and infestations) | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 1
Device related infection (Infections and infestations) | 0 | 0 | 3 | 2
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 1
Empyema (Infections and infestations) | 0 | 1 | 0 | 1
Enterobacter pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 0 | 1 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1
Groin infection (Infections and infestations) | 0 | 0 | 1 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 1
Large intestine infection (Infections and infestations) | 0 | 0 | 1 | 1
Meningitis (Infections and infestations) | 0 | 0 | 1 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Papilloma viral infection (Infections and infestations) | 0 | 0 | 1 | 1
Pleural infection (Infections and infestations) | 0 | 0 | 1 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 17 | 7 | 118 | 137
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 8 | 8
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 2 | 2
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 1 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1 | 3 | 3
Sepsis (Infections and infestations) | 3 | 2 | 22 | 26
Septic shock (Infections and infestations) | 0 | 0 | 3 | 3
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 3 | 4
Urinary tract infection (Infections and infestations) | 1 | 0 | 8 | 9
Urosepsis (Infections and infestations) | 0 | 0 | 2 | 2
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 4
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 4
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 5 | 5
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Product administration error (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 4
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 3 | 3
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 1 | 1
Influenza A virus test positive (Investigations) | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 1
Staphylococcus test positive (Investigations) | 0 | 0 | 1 | 1
Troponin I increased (Investigations) | 0 | 0 | 1 | 1
Troponin increased (Investigations) | 1 | 0 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 33 | 35
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 8 | 8
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 9 | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 8 | 10
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 11 | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 9 | 10
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | 6
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 7 | 7
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 15 | 509 | 521
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 6 | 6
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 9 | 10
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 6 | 6
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 3
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Respiratory papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 1
Central nervous system haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebellar stroke (Nervous system disorders) | 1 | 0 | 1 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 2 | 2
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 9 | 10
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 3 | 3
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 3
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 2 | 3
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 3 | 3
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 0 | 2 | 3
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 2 | 2
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 3 | 3
Lacunar stroke (Nervous system disorders) | 0 | 0 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1 | 2
Seizure (Nervous system disorders) | 2 | 1 | 12 | 14
Spinal cord compression (Nervous system disorders) | 0 | 0 | 9 | 9
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 9 | 11
Vocal cord paralysis (Nervous system disorders) | 1 | 0 | 0 | 1
Device malfunction (Product Issues) | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 2 | 2
Confusional state (Psychiatric disorders) | 1 | 1 | 11 | 12
Delirium (Psychiatric disorders) | 0 | 0 | 3 | 3
Depression (Psychiatric disorders) | 1 | 1 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 9 | 9
Psychotic disorder (Psychiatric disorders) | 2 | 0 | 0 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 15 | 15
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 4 | 4
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal pain (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1
Adnexal torsion (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 18 | 18
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 27 | 31
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 91 | 92
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 10 | 10
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 16 | 17
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 37 | 38
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 23 | 24
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 10 | 10
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 40 | 43
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 22 | 23
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 16 | 17
Embolism (Vascular disorders) | 0 | 1 | 7 | 7
Haematoma (Vascular disorders) | 0 | 1 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 2 | 2
Hypertensive urgency (Vascular disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 7 | 7
Jugular vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 0 | 2 | 2
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 4 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Nivolumab Monotherapy (Post-Randomization) (N=127) | Cohort B: Nivolumab Monotherapy (Post-Randomization) (N=125) | Nivolumab Monotherapy (Pre-Randomized) (N=1428) | Nivolumab Monotherapy (Total) (N=1428)
Anaemia (Blood and lymphatic system disorders) | 11 | 7 | 208 | 222
Hypothyroidism (Endocrine disorders) | 8 | 4 | 129 | 136
Abdominal pain (Gastrointestinal disorders) | 14 | 7 | 117 | 133
Constipation (Gastrointestinal disorders) | 9 | 6 | 274 | 290
Diarrhoea (Gastrointestinal disorders) | 36 | 17 | 275 | 292
Nausea (Gastrointestinal disorders) | 22 | 9 | 332 | 352
Vomiting (Gastrointestinal disorders) | 15 | 5 | 191 | 207
Asthenia (General disorders) | 5 | 0 | 73 | 79
Fatigue (General disorders) | 26 | 17 | 516 | 544
Non-cardiac chest pain (General disorders) | 6 | 3 | 84 | 94
Oedema peripheral (General disorders) | 13 | 9 | 180 | 197
Pyrexia (General disorders) | 16 | 2 | 123 | 143
Bronchitis (Infections and infestations) | 14 | 5 | 50 | 64
Pneumonia (Infections and infestations) | 15 | 14 | 89 | 102
Sinusitis (Infections and infestations) | 8 | 4 | 59 | 65
Upper respiratory tract infection (Infections and infestations) | 28 | 15 | 128 | 153
Urinary tract infection (Infections and infestations) | 12 | 11 | 60 | 75
Fall (Injury, poisoning and procedural complications) | 11 | 10 | 54 | 65
Blood creatinine increased (Investigations) | 17 | 4 | 65 | 76
Weight decreased (Investigations) | 12 | 20 | 182 | 192
Weight increased (Investigations) | 15 | 4 | 39 | 48
Decreased appetite (Metabolism and nutrition disorders) | 18 | 13 | 313 | 336
Dehydration (Metabolism and nutrition disorders) | 9 | 3 | 127 | 134
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 4 | 61 | 68
Hypokalaemia (Metabolism and nutrition disorders) | 16 | 9 | 126 | 138
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 | 8 | 149 | 162
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 5 | 97 | 102
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 18 | 284 | 314
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 11 | 189 | 211
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 4 | 44 | 57
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 8 | 74 | 82
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9 | 2 | 90 | 102
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 6 | 60 | 67
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 44 | 50
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 8 | 101 | 112
Dizziness (Nervous system disorders) | 17 | 7 | 140 | 156
Headache (Nervous system disorders) | 17 | 8 | 140 | 161
Anxiety (Psychiatric disorders) | 7 | 3 | 96 | 106
Depression (Psychiatric disorders) | 3 | 5 | 71 | 75
Insomnia (Psychiatric disorders) | 15 | 7 | 128 | 147
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 12 | 9 | 41 | 54
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 22 | 302 | 331
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 17 | 339 | 359
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | 82 | 88
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 49 | 58
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 51 | 55
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 33 | 42
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 | 7 | 94 | 105
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 21 | 30
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 71 | 80
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 5 | 119 | 127
Rash (Skin and subcutaneous tissue disorders) | 10 | 5 | 98 | 108
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 | 4 | 62 | 72
Rash pruritic (Skin and subcutaneous tissue disorders) | 7 | 0 | 37 | 42
Hypertension (Vascular disorders) | 12 | 6 | 56 | 64
Hypotension (Vascular disorders) | 7 | 5 | 70 | 79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT02066636/Prot_SAP_000.pdf